CLINICAL TRIAL: NCT00793156
Title: A Randomized-Withdrawal Phase 3 Study Evaluation the Safety and Efficacy of Oral Nalfurafine HCl (AC-820)in Subjects on Hemodialysis With Uremic Pruritus (Renal Itch)
Brief Title: A Randomized-Withdrawal Phase 3 Study Evaluating the Safety and Efficacy of Oral Nalfurafine HCl (AC-820)in Subjects on Hemodialysis With Uremic Pruritus (Renal Itch)
Acronym: AC120-8231
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Acologix, Inc. (Industry)
Responsible Party: Dawn McGuire, MD, Acologix, Inc
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: AC120-8231
Record Dates: First submitted 2008-11-17; First posted 2008-11-19 (Estimated); Last update posted 2010-02-04 (Estimated); Status verified 2010-02

CONDITIONS: Uremic Pruritus
Keywords: uremic pruritus

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Placebo (Placebo Comparator): Patients will be randomized into Placebo group
  Interventions: Other: Placebo
- 2 (Active Comparator): 2.5 µg group randomized
  Interventions: Drug: Nalfurafine HCl 2.5 µg
- 3 (Active Comparator): 5.0 µg group randomized
  Interventions: Drug: Nalfurafine HCl 5.0 µg

INTERVENTIONS:
Drug: Nalfurafine HCl 2.5 µg — Daily dose of 2.5 µg
  Arms: 2
Drug: Nalfurafine HCl 5.0 µg — Daily dose of 5.0 µg
  Arms: 3
Other: Placebo — Placebo daily dose
  Arms: Placebo

SUMMARY:
Primary objective of this multicenter, double-blind, placebo controlled, randomized withdrawal study are to determine the effectiveness and safety of orally administered AC-820 in doses of 2.5 µg and 5.0 µg daily in patients with moderate to severe itching associated with end-stage renal disease and hemodialysis, and perform a population PK analysis.

ELIGIBILITY:
Inclusion Criteria:

* 18 yrs old or older
* moderate to severe pruritus
* end stage renal disease
* 3x weekly hemodialysis

Exclusion Criteria:

* pruritus not due to renal disease
* abnormal liver function
* Ca-P > 80 mg/dl or HgB <8.5 g/dl or PTH > pg/mL
* Within four months spKt/V < 1.05

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 350 (Estimated)
Dates: Start 2009-12; Primary Completion 2010-12 (Estimated); Study Completion 2011-03 (Estimated)

PRIMARY OUTCOMES:
Primary efficacy endpoint is the change in worst itching intensity from baseline, compared to that in the last two weeks of the double blind, placebo controlled, randomized withdrawal period. | 11 weeks

REFERENCES:
- [Derived] Hercz D, Jiang SH, Webster AC. Interventions for itch in people with advanced chronic kidney disease. Cochrane Database Syst Rev. 2020 Dec 7;12(12):CD011393. doi: 10.1002/14651858.CD011393.pub2. PMID 33283264